CLINICAL TRIAL: NCT00463632
Title: Schistosomiasis in Women of Reproductive Age in Burkina Faso: Implications for Control
Status: Completed | Type: Observational
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Centre Muraz (Other)
Other Study IDs: SRP-BF-ST-06
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Schistosomiasis; Anaemia; Pregnancy
Keywords: schistosomiasis; anaemia; pregnancy
MeSH Terms: conditions — Schistosomiasis; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — urine faeces blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Cross-sectional study of prevalence and intensity of schistosome infection in pregnant women, follow-up into postpartum, and the association of schistosome infection with haemoglobin concentration, compared to a group of non-pregnant women.

DETAILED DESCRIPTION:
The objective of this study is to investigate the epidemiology of schistosomiasis and anaemia among pregnant and non-pregnant women in Burkina Faso and explore the implications for the national schistosomiasis control programme and future studies.

Specific objectives are:

* to determine the prevalence and intensity of schistosome infection in pregnant women attending for antenatal care and in non-pregnant women of reproductive age in an area which is hyperendemic for S.haematobium infection and in which there is little or no S.mansoni infection
* to determine the prevalence and intensity of schistosome infection in pregnant women attending for antenatal care and in non-pregnant women of reproductive age in an area in which S.mansoni infection is common
* to determine Haemoglobin concentration in pregnant women attending for antenatal care and in non-pregnant women of reproductive age in the regions described above
* to investigate the association between infection and haemoglobin concentration in pregnant and non-pregnant women
* to determine the prevalence of other parasitic infections in pregnant women and non-pregnant women including hookworms, ascaris, trichuris and malaria
* to demonstrate the research team's ability to follow-up pregnant women recruited at antenatal care clinics onto the postpartum period

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending for ANC
* Non-pregnant women age 15-45 years accompanying relatives or children to the health centres or for immunization

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: antenatal care clinics child immunization program
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seydou Touré, MD, Principal Investigator — The National Schistosomiasis Control Program Burkina Faso
Locations (2):
- Burkina Faso (2):
  - Dori Health Centre, Dori
  - National Schistosomiasis Control Program, Ouagadougou